CLINICAL TRIAL: NCT00870935
Title: A Prospective, Randomized Study to Compare the Efficacy and the Tolerability of Three Methods of Performing Hysterosalpingography
Brief Title: A Trial to Compare Three Methods of Performing Hysterosalpingography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Giuseppe Ricci, IRCCS Burlo Garofolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RU02/07
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2009-03

CONDITIONS: Infertility
Keywords: Balloon catheter; Cervical vacuum cup; Hysterosalpingography; Infertility; Pain; Fallopian Tube Patency Tests; Female Infertility
MeSH Terms: conditions — Infertility; Pain; Infertility, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Balloon catheter (Active Comparator): Hysterosalpingography using intrauterine Balloon catheter
  Interventions: Procedure: Balloon catheter
- Cervical vacuum cup (Active Comparator): Hysterosalpingography using cervical vacuum cup
  Interventions: Procedure: Cervical vacuum cup
- Operator choice (Experimental): Hysterosalpingography is performed using either balloon catheter or cervical vacuum cup on the basis of the operator's choice
  Interventions: Procedure: Balloon catheter; Procedure: Cervical vacuum cup

INTERVENTIONS:
Procedure: Balloon catheter — Hysterosalpingography is performed using intrauterine balloon catheter
  Arms: Balloon catheter; Operator choice
Procedure: Cervical vacuum cup — Hysterosalpingography is performed using cervical vacuum cup
  Arms: Cervical vacuum cup; Operator choice

SUMMARY:
The purpose of this study is:

* to determine whether the choice of the device for performing hysterosalpingography on the basis of the cervix characteristics can reduce the procedure failure rate;
* to determine whether patient medical history is correlated with the degree of pain experienced during the HSG procedure.

DETAILED DESCRIPTION:
A group of women will be randomized to undergo HSG, using 1) a balloon catheter in a first group of patients; 2) a cervical vacuum cup in a second group; 3) one of the two devices decided by the operator depending on the cervix characteristics in a third group (that will be named "operator's choice").

The operator will ask the woman to evaluate the degree of pain experienced during the application of the device and the injection of the contrast, after 2, 6 and 24 hours. The degree of pain will be evaluated using the VAS system, an analogue scale rating from 1 to 10.

A nurse will notice the patient's reaction and will evaluate the pain, depending on the movements of the hands and the body and the woman's moaning. Moreover, the assistant will note down the personal data and the history of the patient. The operator will record the objective and subjective difficulty of the performance, using a rating scale from 0 to 9. The length of the procedure, the volume of contrast used, the amount of radiations and the time of exposure of the patient will also be considered.

At the end of HSG both the gynaecologist and the radiologist will express their satisfaction upon the examination with a score from 0 to 10.

ELIGIBILITY:
Inclusion Criteria:

* infertility

Exclusion Criteria:

* hypersensitivity to iodine or radio-opaque contrast dye
* cervicitis
* genital bleeding
* genital malignancy

Ages: 25 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 222 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
failure rate to complete hysterosalpingography (HSG) | two years

SECONDARY OUTCOMES:
the objective difficulty to perform HSG | two years
the subjective difficulty to perform HSG | two years
the fluoroscopic time | two years
the length of the procedure of device application | two years
the volume of contrast medium used | two years
gynecologist satisfaction with the procedure | two years
radiologist satisfaction with the procedure | two years
the percentage of short-term complications | two years
the percentage of long-term complications | two years
correlation between patient medical history and the degree of pain experienced during the HSG procedure | two years
the degree of pain experienced during the HSG procedure | two years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Ricci, MD, Principal Investigator — IRCCS Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy